CLINICAL TRIAL: NCT03882697
Title: Ability of Cardio Q for Prediction of Hypotension After Postural Change in Robot-Assisted Laparoscopic Radical Prostatectomy
Brief Title: Ability of Cardio Q for Prediction of Hypotension
Status: Completed | Type: Observational
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Associate professor, Severance Hospital
Other Study IDs: 4-2018-0976
Record Dates: First submitted 2019-02-12; First posted 2019-03-20 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
Keywords: Robotic surgery; Position; Cardio Q; hypotension
MeSH Terms: conditions — Prostatic Neoplasms; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation the ability of each indicator of Cardio Q in predicting hypotension after position changes in robot-assisted laparoscopic radical prostatectomy

DETAILED DESCRIPTION:
Hypotension is common in patients who undergo general anesthesia. Hypotension may cause hypoperfusion in the organs of the body, resulting in ischemia and increased mortality within one year. Hypotension may occur at any time during general anesthesia but may also occur with changes in posture. In robot-assisted laparoscopic radical prostatectomy, hypotension often occurs when posture is changed from a Trendelenburg position to a supine position. However there is no data regarding which hemodynamic parameters can predict hypotension induced by position change.

Excessive administration of the fluid in steep Trendelenburg position may lead to fluid overload and lead to complications such as pulmonary edema. Thus, the predictors are should be identified to manage patients without fluid overload. Therefore, the aim of this study is to investigate the parameters of Cardio Q which are useful for predicting hypotension after position change.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing robot-assisted laparoscopic radical prostatectomy ASA 1-3

Exclusion Criteria:

Patients that

* Unstable angina, left ventricular ejection fraction <40%
* Severe vascular disease
* Insertion type : pacemaker / defibrillator
* Autonomic nervous system diseases
* When esophageal varices are present
* If the subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male can have prostate
Study Population: ASA 1-3 Patient undergoing robot-assisted laparoscopic radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | Before position change, After position change (1, 3, 5, 7, and 10 minutes)
  The changes mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (2):
- South Korea (2):
  - Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Severance Hospital, Yonsei University College of Medicine, Seoul
  - Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim NY, Kim KJ, Kim TL, Shin HJ, Oh C, Lee MH, Min JY, Kim SY. Prediction of hypotension after postural change in robot-assisted laparoscopic prostatectomy using esophageal Doppler monitoring: a prospective observational trial. Sci Rep. 2021 Jul 16;11(1):14589. doi: 10.1038/s41598-021-93990-3. PMID 34272425